CLINICAL TRIAL: NCT01447485
Title: A Multicenter, Open-label, Single-dose Study to Evaluate the Pharmacokinetics of Valsartan in Japanese Pediatric Patients 6 to 14 Years of Age
Brief Title: Pharmacokinetics Following Single-dose of Valsartan in Japanese Pediatric Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CVAL489K1101
Record Dates: First submitted 2011-08-31; First posted 2011-10-06 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2012-05

CONDITIONS: Hypertension; Chronic Kidney Disease; Nephrotic Syndrome
Keywords: Hypertension, chronic kidney disease; nephrotic syndrome; pharmacokinetics
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Nephrotic Syndrome | interventions — Valsartan

ARMS (1):
- Valsartan 20 mg or 40 mg (Experimental)
  Interventions: Drug: Valsartan (VAL489)

INTERVENTIONS:
Drug: Valsartan (VAL489)

SUMMARY:
This study will assess the pharmacokinetics and safety following single dose of valsartan in Japanese pediatric patients with hypertension, chronic kidney disease, or nephrotic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Japanese pediatric patients with hypertension, chronic kidney disease, or nephrotic syndrome

Exclusion Criteria:

* GFR < 30 mL/min/1.73 m2
* Inability to safely tolerate the temporary discontinuation of concomitant antihypertensive medications (expect amlodipine or atenolol) from 24 hours prior to study drug administration to study completion.
* Inability to safely tolerate the temporary discontinuation of any drug known or suspected to effect hepatic or renal clearance capacity from 24 hours prior to study drug administration to study completion (this includes drugs that are known to cause induction or inhibition of hepatic enzymes).

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
AUC of valsartan in plasma | Up to 24 hours post-dose
Cmax of valsartan in plasma | Up to 24 hours post-dose
Tmax of valsartan in plasma | Up to 24 hours post-dose
T1/2 of valsartan in plasma | Up to 24 hours post-dose
CL/F of valsartan in plasma | Up to 24 hours post-dose

SECONDARY OUTCOMES:
ECG evaluations | 24 hours post-dose
Standard clinical laboratory evaluations | 24 hours post-dose
Vital signs | 2, 4, and 24 hours post-dose
Physical examination | 24 hours post-dose
Number and severity of adverse events | Up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Tokyo

REFERENCES:
- See also: Results for CVAL489K1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6883